CLINICAL TRIAL: NCT04098757
Title: Observation of Patients Affected by Fibromyalgic Syndrome (FMS): Comparison of Different Therapeutic Approaches
Brief Title: Fibromyalgia Different Approaches: Acupuncture vs Migratens
Acronym: FrIDAy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Vittorio Schweiger (Other)
Responsible Party: Sponsor-Investigator, Vittorio Schweiger, PROFESSOR, Azienda Ospedaliera Universitaria Integrata Verona
Organization: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Other Study IDs: 1917CESC FrIDAy
Record Dates: First submitted 2019-02-18; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Fibromyalgia, Primary; Fibromyalgic Sindrome
Keywords: Fibromyalgia; Fibromyalgic Sindrome (FMS); Pain; Acupuncture; Nutraceutical products
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Migratens: 2 sachets/day: 800 mg of α-Lipoic acid, 450 mg of magnesium bisglycinate, 300 mg of L-Tryptophan, 20 mcg of Vitamin D3, 2.4 mg of Vitamin B2, 25 mg of Niacin, 150 mg of Coenzyme Q10. Patients who receive Migratens food supplementation have to take 2 sachets / day for 12 weeks. The supplement will be prescribed as usual and the assumption of the same will be recorded by partecipants in the appropriate daily; if the subject does not continue the indication the data collected up to that moment will be considered.
  Interventions: Dietary Supplement: Migratens
- acupuncture: 2 sessions a week, for a total of 10 (5 weeks), performed by the same operator, repeatable if necessary, after a therapeutic interval of at least one month. Each session lasts about 20-30 minutes per patient. Tewa J Type sterile disposable needles, coated, with a Chinese-style copper wire handle, with a guide tube, of 22x13 mm (CJ 2213) and 30x25 mm (CJ 3025) will be used. Acupuncture will be carried out by same trained operator.

INTERVENTIONS:
Dietary Supplement: Migratens — 2 sachets/day: 800 mg of α-Lipoic acid, 450 mg of magnesium bisglycinate, 300 mg of L-Tryptophan, 20 mcg of Vitamin D3, 2.4 mg of Vitamin B2, 25 mg of Niacin, 150 mg of Coenzyme Q10. Patients who receive Migratens food supplementation have to take 2 sachets / day for 12 weeks. The supplement will be prescribed as usual and the assumption of the same will be recorded by partecipants in the appropriate daily; if the subject does not continue the indication the data collected up to that moment will be considered.
  Groups: Migratens

SUMMARY:
Fibromyalgia or Fibromyalgic Sindrome (FMS) is a chronic debilitating pain syndrome, characterized by widespread chronic musculoskeletal pain and generalized painful hypersensitivity, which may be associated with systemic, cognitive and psycho-emotional somatic disorders. Etiology is not completely known. The diagnosis of fibromyalgia is anamnestic and clinical, without evident alterations at the objective examination or at laboratory and radiology investigations. According last guidelines, the best approach to treat FMS must be personalized and multidisciplinary, including pharmacological and non-pharmacological interventions. Moreover, a correct treatment of comorbidities, practice of bland physical activity or meditative discipline, as well as a pychological support are very important in FMS.

The aim of this study is to evaluate the activity of some common therapeutic pathways available for FMS: acupuncture and nutraceutical products; the latter are numerous on the market and based on powerful antioxidants. In this case Migratens was chosen for its composition: α-lipoic acid, polyvitaminic complexes (B and D group vitamins), coenzyme Q10, magnesium and tryptophan.

DETAILED DESCRIPTION:
Fibromyalgia or Fibromyalgic Sindrome (FMS) is a chronic debilitating pain syndrome, affecting about 2-4% of the general population, with an average peak between 30 and 50 years, but with a significantly higher prevalence, until about 8-10%, if considered only female sex or greater age. Fibromyalgia is characterized by the presence of widespread chronic musculoskeletal pain and generalized painful hypersensitivity, which may be associated with systemic, cognitive and psycho-emotional somatic disorders, such as: asthenia, sleep disorders, depression, anxiety, headache, paresthesia, dry eye, tachycardia, intercostal pain, dyspnoea, gastrointestinal or gynecological or urological disorders.

Etiology is not completely known, even if genetic, environmental, physical and emotional factors seem to interact and promote an hypersensitive state, both at central and peripheral level, leading to a functional disorder of pain modulation system. Sleep or immune system disorders, focal tissue abnormalities, physical or psychological trauma seem to trigger the disease, but many patients are not able to identify any apparent cause.

Validated questionnaires, including the Fibromyalgia Impact Questionnaire (FIQ), are used to assess the impact of fibromyalgia on people's health and quality of life; in 2016 this survey was revised (FIQR) to intercept almost the entire spectrum (domains) of problems related to the disease and response to treatment, as well as to include other relevant parameters in the evaluation of the FMS patient (eg assessment of cognitive functions, balance problems, etc.), absent in the original version. In this scale the score of each item ranges from 0 to 10. First block of questions concerns the physical function of the subject and the related physical difficulties experienced in the last week; the subtotal score of first 9 items is divided by three, therefore the maximum score is 30. Second domain concerns FMS impact on general health in the last week and consists of two questions; the relative score remains unchanged, so maximum score is 20. Third domain consists of 10 items concerning the severity of main symptoms related to fibromyalgia experienced in the last week; addition of these is divided by two, thus maximum score is 50. Sum of all three domains corresponds to the total of the questionnaire and its interpretation is as follows: 0-42 mild FMS, 43-59 moderate FMS, 60-74 severe FMS, 75-100 FMS very serious. In this survey also depression is valuated, in a scale from 0 (absence of mood disorder) to 10 (severe depression).

Visual Analogue Scale (VAS) is a visual representation of severity of pain felt by the patient, indicated on a 10 cm long line, where one end indicates the absence of ache (0), while the other corresponds to the worst pain imaginable (10).

According last guidelines, the best approach to treat FMS must be personalized and multidisciplinary, including pharmacological and non-pharmacological interventions. Drugs, with off-label indication for fibromyalgia, are amitriptyline, duloxetine and pregabalin, in monotherapy or combined. If there is no response, patients may try to employ analgesics and anti-inflammatories as needed or use complementary and alternative therapies (for example: acupuncture, transcranial stimulation or TENS, cannabinoid derivatives, nutraceutical products, vitamin D supplementation). Moreover, a correct treatment of comorbidities, practice of bland physical activity or meditative discipline, as well as a pychological support are very important in FMS.

The aim of this study is to evaluate the activity of some common therapeutic pathways available for FMS: acupuncture and nutraceutical products. The first one involves treating the most painful areas with local, adjacent and distant points, as well as treating basic condition, framed according to Traditional Chinese Medicine (TCM). In clinical practice, selection of acupoints must be based on diagnostic criteria of TCM and aimed to reduce symptoms, therefore it must be personalized as much as possible, even if some points of treatment are more frequent. Metal needles, placed into specific acupoints, modulate the release of various pain neuromediators (serotonin, substance P, neuro peptide Y, endorphins), in addition to activate a local and systemic anti-inflammatory effect, with further sedative properties on pain. Moreover, there are evidences that acupuncture enhances the effect of pharmacological treatment (antidepressants) and exercise on pain reduction of 30% (30 points on a pain scale from 0 to 100), with almost null adverse effects.

Numerous nutraceutical products for fibromyalgia are available on the market; among these Migratens was chosen for its composition: in fact it contains α-lipoic acid, a powerful endogenous antioxidants, polyvitaminic complexes (B and D group vitamins) and coenzyme Q10, essential for correct cellular functionality, magnesium and tryptophan, mineral and essential aminoacid with positive effects on skeletal muscle system, sleep and mood disorders.

This study expects to evaluate which of these treatment, acupuncture and nutraceutical products, allow a pain reduction, but also an improvement of general well-being, with positive effects on somatic or psycho-emotional symptoms, without significant side effects added.

WPI, SSS, Fibromyalgia Impact Questionnaire-Revised (FIQR), Visual Analogic Scale are instrument to estimate FMS severity at different time: at the fist patient evaluation, during treatment time and at the end of the study, after at least three month free from therapy.

Sixty-one female fibromyalgic patients were recruited for this study and randomized for the two possible treatments: 27 of them were assigned to Group A, for a therapy of three months with Migratens (2 sachets/day), and 34 to Group B, treated with ten (one cycle) or twenty (two cycles, with a month break between cycles) acupuncture sessions, carried out by the same operator. The subjects assigned to the two groups follow the normal controls, during which the participants have to indicate number, type and dosage of the symptomatic drugs taken in a daily allowance. Another check will also be performed at six months from the beginning of enrollment, after at least three months free of treatment. In fact, it is interesting to understand which therapeutic strategy is most effective and which one presents a more lasting pain reduction over time from the end of treatment to the subsequent follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients not under pharmacological treatment for at least six months,
* patients with a new diagnosis of fibromyalgia (FM)
* hypovitaminosis D (vitamin D <30 mg / ml) or patients already in oral supplementation with 1,000 IU / day. People with hypovitaminosis are treated with Vitamin D supplementation
* 30 - 65 years old
* female sex
* signature of informed consent

Exclusion Criteria:

* patients treated with active drugs on the neuroendocrine system
* intake of drugs that can influence skeletal metabolism
* addition of other fibromyalgia medicines other than those included in the study, during the observational period
* allergies to components of the food supplement used
* use of oral hypoglycemic agents
* participation in other studies
* recent acupuncture treatments elsewhere
* severe psychiatric or neurological disorders

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female affected by fybromialgia age between 30-65 years old
Study Population: Patients suffering from fibromyalgia for at least 6 months according to the modified criteria of 2016 affering to Verona's Hospital
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale pain reduction in fibromyalgic patients from baseline to 6 months follow-up | 6 months
  to observe pain reduction in fibromyalgic patients treated with nutraceutic (Migratens®) - Groupo A, and with acupuncture - Group B, at the end of the study. visual analogue scale is anagogic scale that evaluate continuous aspect of the scale differentiates it from discrete scales such as the Likert scale, from 0 to 10.

SECONDARY OUTCOMES:
visual analogue scale pain reduction in fibromyalgic patients from baseline to 1 month follow-up, from baseline to 3 months follow-up | 1 and 3 months
  - to observe pain reduction in fibromyalgic patients treated with nutraceutic (Migratens®) - Groupo A, and with acupuncture - Group B, at different follow up time visual analogue scale is anagogic scale that evaluate continuous aspect of the scale differentiates it from discrete scales such as the Likert scale, from 0 to 10.
Cenestesi improvement measured with revised Fibromyalgia Impact Questionnaire SCORE in fibromyalgic patients from baseline to 6 months follow-up | 6 months
  to value general improvement of cenestesi between two groups. each of the 9 questiona of questionnaire present a score from 0 to 10 to evaluate haw fibromyalgia make activities difficult, zero score correspond to no difficult and 10 to always difficult.
visual analogue scale pain reduction in fibromyalgic patients from 3 month to 6 month | 3 and 6 months
  to observe time of pain reduction or pain free after treatment end. visual analogue scale is anagogic scale that evaluate continuous aspect of the scale differentiates it from discrete scales such as the Likert scale, from 0 to 10.
percentage of adverse effect | 6 months
  to observe number and type of treatment adverse effect during study time

CONTACTS AND LOCATIONS:
Locations (1):
- Nrc, Verona, Italia, Italy

IPD SHARING:
Plan to Share IPD: No